CLINICAL TRIAL: NCT02827552
Title: Integrative Molecular Analysis of Individual Radiosensitivity Among a Population of Pediatric Patients Treated With Radiation in Eastern France.
Brief Title: Description of Individual Radiosensitivity With Molecular Biomarkers in a Pediatric Oncology Population
Acronym: ARPEGE BioM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The liquidation of our industrial partner NEOLYS Diagnostics, directly involved in the methodology of the study and a sub-optimal rate of inclusions which did not allow us to include all patient within the allotted time.
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00975-44
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Cancer-related Problem/Condition
Keywords: pediatric oncology; radiotherapy; radiosensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARPEGE BioM (Other): N/A (not a randomized study)
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy — skin biopsy performed prior radiation to characterize in blind the individual radiosensitivity of the patient

SUMMARY:
This study aims to explore prospectively the distribution of individual radiosensitivity in the pediatric population and to determine the predictive power of individual radiosensitivity biomarkers from an immunofluorescence technique on primary dermal fibroblasts

DETAILED DESCRIPTION:
900 children and adolescents benefit from radiation each year in France. The mean age at diagnosis is 5 years; life expectancy for the 80% of them who could cure is long, and the incidence of radiation-related acute and mainly late complications - not evaluated to date - could exceed that of adults. Dysfunction of irradiated organs and growth disorders are specific to the pediatric subpopulation. Individual radiosensitivity of children and adolescents is unknown at this time, probably with large variability depending on the age when considering the changes in metabolic functions throughout growth. These complications are largely attributable to inter individual constitutional variations of cellular response to DNA damage.

Subject to radiation-induced DNA damages such as double-strand breaks (DSB), cells reacts by triggering a whole series of phosphorylation events coordinated within multi protein complexes whose interplay is still misknown (DNA damage response i.e. DDR). Indirect Immunofluorescence cell scanning has revolutionized radiation biology research by permitting the detection of individual DSB in each cell nucleus in a dose range from 1 mGy to 10 Gy. This technique has notably confirmed that yield of unrepaired DSB is correlated with cell RS. From a broad spectrum of human radiosensitive skin fibroblast cell lines, the Inserm CRU 1052 team proposed a general model of DSB signaling and repair and a molecular assay to stratify patients according to their individual RS.

ARPEGE biomarqueurs is a prospective multicenter study to prospectively evaluate with this assay the RS of children and adolescents treated over a year in all pediatric oncology departments of the Region Grand Est and set thresholds in this population. 150 children are thus potentially includable in different centers. The assay will be performed on primary fibroblasts cultured from a skin biopsy taken at diagnosis. The RS of patients will be measured in blind. Confusion factors such as irradiated volume, skin phototype, previous chemotherapy regimen, smoking, comorbities (diabetes, immunodeficiency, chronic inflammatory disease ...) will be reported. In parallel the RT-acute toxicity will be reported according to NCI-CTCAE v4.0 reference scale three months of the completion of RT then periodically during 15 years.

Screening hypersensitive patients would be a major step forward in the management of cancers, opening a view to personalized medicine.

ELIGIBILITY:
Inclusion Criteria:

* Children < 18 years old
* Patient with an indication of radiotherapy
* Patient must be affiliated to a social security system
* Patient under parental autority
* Ability to provide an informed written consent form

Exclusion Criteria:

* Contraindications for skin biopsy
* Contraindications for radiotherapy
* Referred to palliative radiotherapy
* Prior radiotherapy in the same area
* Indication of hypofractionated radiotherapy
* Patient monitoring impossible
* Patients deprived of liberty or under supervision

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
skin fibroblast radiosenstivity | up to 5 months
  residual double-strand breaks 24h after ex vivo radiation assessed with indirect immunofluorescence (gammaH2AX marker).

SECONDARY OUTCOMES:
early cutaneous, mucosal and hematological early radiation toxicity | 3 months
  early radiation toxicity pattern assessed according to CTACAE v4.0 scale
pATM nucleoshuttling | up to 5 months
  pATM foci counted 10 minutes and 1 hour after ex vivo radiation assessed with indirect immunofluorescence (pATM marker).
mean micronuclei number | up to 5 months
  micronuclei counted 24 hours after ex vivo radiation assessed with indirect immunofluorescence (DAPI marker).
late radiation toxicity | 15 years
  deterministic tissue effects as well as secondary malignancies occurring in radiation field more than 3 months and up to 15 years after RT, using CTCAE v4.0 scale

CONTACTS AND LOCATIONS:
Overall Officials: VOGIN GUILLAUME, MD,PhD, Principal Investigator — Institut de Cancérologie de Lorraine; BERNIER CHASTAGNER VALERIE, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (11):
- France (11):
  - CHU de Besançon, Besançon
  - CHU de Dijon, Dijon
  - Georges-François-Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - CHU de Reims, Reims
  - Centre Paul Strauss, Strasbourg
  - Hôpital de Hautepierre, Strasbourg
  - CHRU toulouse, Toulouse
  - IUCT Oncopole, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - CHRU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernier-Chastagner V, Hettal L, Gillon V, Fernandes L, Huin-Schohn C, Vazel M, Tosti P, Salleron J, Francois A, Cerimele E, Perreira S, Peiffert D, Chastagner P, Vogin G. Validation of a high performance functional assay for individual radiosensitivity in pediatric oncology: a prospective cohort study (ARPEGE). BMC Cancer. 2018 Jul 6;18(1):719. doi: 10.1186/s12885-018-4652-7. PMID 29976172